CLINICAL TRIAL: NCT02547584
Title: Impact of Anxiety on Cardiac Substrate Modification in Women With Atrial Fibrillation Undergoing Catheter Ablation
Acronym: AWARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive Medical Director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCAI_AWARE
Record Dates: First submitted 2015-09-03; First posted 2015-09-11 (Estimated); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: with baseline anxiety+catheter ablation (Active Comparator): Baseline anxiety will be defined as; Cardiac Anxiety Questionnaire (CAQ) score >2.14 Hospital Anxiety and Depression Questionnaire (HAD) >7 State-Trait Anxiety Inventory (STAI): State-anxiety score >40
  Interventions: Procedure: Catheter ablation
- Group 2: Without baseline anxiety + catheter ablation (Active Comparator): Cardiac Anxiety Questionnaire (CAQ) score <2.14 Hospital Anxiety and Depression Questionnaire (HAD) <7 State-Trait Anxiety Inventory (STAI): State-anxiety score <40
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — Pulmonary vein antrum isolation (PVAI) plus entire posterior wall plus coronary sinus plus left part of the septum. This intervention will be received by all as standard of care
  Other Names: RFCA

SUMMARY:
This pilot study aims to assess the impact of anxiety on the cardiac substrate remodeling in female patients with paroxysmal and persistent atrial fibrillation (AF).

DETAILED DESCRIPTION:
Hypothesis: High level of anxiety promotes remodeling of cardiac substrate via persistent inflammation, resulting in an increase in the prevalence of left atrial scar and non-pulmonary vein (non-PV) triggers in women with AF.

Rationale: Anxiety is generally defined as a psycho-biological emotional state or reaction that consists of unpleasant feelings of tension, apprehension, nervousness, and worry, and activation of the autonomic nervous system. This disorder is typically more common in women than men. There is considerable evidence to suggest close interactions between anxiety and inflammation and inflammation and AF.

Earlier studies have documented strong association between anxiety and inflammation as shown by high levels of inflammatory biomarkers such as C-reactive protein (CRP), total white blood cell (TWBC) count, fibrinogen and interleukin-6 in patients with anxiety. Chronic inflammation results in structural remodeling of the atrial architecture such as fibrotic changes that supports genesis and perpetuation of AF. In cardiac fibrosis, myocytes coupled with fibroblasts can undergo early depolarization resulting in increased ectopic beats and repetitive firing leading to the origin of non-pulmonary vein (non-PV) drivers. Left atrial scar is another known consequence of cardiac fibrosis. Therefore, it is prudent to hypothesize that high level of anxiety for prolonged period results in structural remodeling of cardiac substrates evidenced by increased prevalence of left atrial scar and non-PV triggers in female patients with paroxysmal and persistent AF.

Scar and non-PV triggers are known independent predictors of arrhythmia recurrence in AF patients undergoing catheter ablation. Recurrences of AF, despite complete PV disconnection, strongly suggest an important possible role of these foci in serving as a source for the persistence of this arrhythmia. Altered conduction and barriers resulting from the atrial scar form the critical circuits for intra-atrial re-entry that promotes AF persistence.

Recent progress in technology and knowledge have provided better understanding and allowed the electrophysiologists to improve on the ablation procedure in order to make it more safe and effective. However, there are still scores of unanswered questions in this relatively young research domain, one of which is if anxiety impacts cardiac substrate remodeling that potentially influences ablation-outcome. Also, of note, anxiety affects how patients perceive their illness, particularly for women, and influence healthcare utilization and economic burden. Therefore, if the role of anxiety would be ascertained, timely intervention of the same would lead to improvement in the success rate of the ablation therapy in females that highly dominate this subset of AF population.

Study Design: This pilot study will prospectively enroll 152 consenting female patients undergoing catheter ablation for AF. Eligible patients will be enrolled after signing informed consent, approved by Institutional Review Board of the participating institution.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years
2. Sex: female
3. Undergoing catheter ablation for paroxysmal or persistent AF
4. Able and willing to provide written informed consent

Exclusion Criteria:

1. Receiving behavioral therapy or medications for the anxiety disorder
2. On hormonal supplement
3. On long-term steroid or anti-inflammatory drugs

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between baseline anxiety score and prevalence of left atrial scar and non-pulmonary vein triggers | intraoperative

SECONDARY OUTCOMES:
Correlation of baseline anxiety score with scar severity | intraoperative
Correlation of baseline TWBC and CRP level with the anxiety score | baseline
Change in CAQ score | 12 months
Recurrence status | 1 year
  Recurrence of AF/ AFlutter/ atrial tachycardia off or on anti-arrhythmic drugs
Change in HAD score | 12 months
Change in State-anxiety | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mitra Mohanty, MD MS FHRS, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (1):
- Texas Cardiac Arrhythmia Institute, St. david's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No